CLINICAL TRIAL: NCT03006432
Title: ESSAI DE PHASE III RANDOMISE EVALUANT LE FOLFOX AVEC OU SANS DOCETAXEL (TFOX) EN 1ère LIGNE DE CHIMIOTHERAPIE DES ADENOCARCINOMES OESO-GASTRIQUES LOCALEMENT AVANCES OU METASTATIQUES
Brief Title: PHASE III RANDOMISED TRIAL to EVALUATE FOLFOX with or WITHOUT DOCETAXEL (TFOX) AS 1st LINE CHEMOTHERAPY for LOCALLY ADVANCED or METASTATIC OESOPHAGO-GASTRIC CARCINOMA
Acronym: GASTFOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: UNICANCER (Other); GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 51
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: OESOPHAGO-GASTRIC CARCINOMA
Keywords: OESOPHAGO-GASTRIC CARCINOMA
MeSH Terms: interventions — Oxaliplatin; Docetaxel; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFOX (Active Comparator): Cycles every 15 days until progression desease
  Interventions: Drug: Oxaliplatin; Drug: 5Fluorouracil bolus; Drug: 5Fluorouracil continu; Drug: Folinic Acid
- TFOX (Experimental): Cycles every 15 days until progression desease
  Interventions: Drug: Oxaliplatin; Drug: 5Fluorouracil continu; Drug: Docetaxel; Drug: Folinic Acid

INTERVENTIONS:
Drug: Oxaliplatin
Drug: 5Fluorouracil bolus
  Arms: FOLFOX
Drug: 5Fluorouracil continu
Drug: Docetaxel
  Arms: TFOX
Drug: Folinic Acid

SUMMARY:
Gastric cancer is the fourth commonest cancer and the second largest cause of mortality from cancer. Surgical resection of localised forms of gastric cancer offers the only chance of a cure. The vast majority of patients, however, present with advanced disease from the outset (locally advanced or metastatic) or recurrent after resection of a localised form.

For metastatic or locally advanced stages of gastric or gastro-oesophageal junction adenocarcinoma, the combination of 2 chemotherapy drugs (dual therapy) as compared with monotherapy or no chemotherapy, makes it possible to improve the tumour response and patient survival. Dual therapy comprising cisplatin + fluoropyrimidine (CF protocol) is considered as one of the first-line chemotherapy treatment standards.

The addition of docetaxel to the CF regime (referred to as the DCF protocol) has made it possible to improve the tumour response rate, the time to tumour progression and overall survival in a randomised phase III trial. This improvement in treatment efficacy was achieved, however, at the expense of a significant increase in grade 3-4 toxicity, including diarrhoea , neutropenia, and neutropenia with complications. Although DCF is considered as a therapeutic standard for advanced forms of gastric cancer, its use is limited in clinical practice due to its high toxicity.

Oxaliplatin has shown its usefulness in treatment of oesophagogastric cancer, with an efficacy at least equal to that of cisplatin. Peripheral sensory neuropathy was less common in the 5FU-cisplatin arm. In terms of treatment efficacy, 5FU-oxaliplatin versus 5FU-cisplatin was associated with a non-significant improvement in median progression free survival rates, and overall survival.

All these data thus suggest that 5FU-oxaliplatin is at least as efficacious and is better tolerated than 5FU-cisplatin, and also that docetaxel-5FU-cisplatin is more efficacious than 5FU-cisplatin, with limited use due to its high toxicity. In the logical continuation of development of chemotherapy protocols for metastatic gastric cancer, the question therefore arises of the usefulness of adding docetaxel to 5FU-oxaliplatin, in terms of efficacy and also tolerance.

In France, chemotherapy with FOLFOX is used extensively as a first line of treatment in advanced gastric cancer, but with progression-free survival and median survival rates that are still too low, and a poor response rate. The use of docetaxel at a dose of 50 mg/m2 every 2 weeks in combination with FOLFOX (TFOX protocol) has shown very interesting results in phase II studies in terms of efficacy and tolerability, and these are worth confirming through a phase III randomised trial. In fact, if these results are confirmed in phase III, TFOX could become the new first-line therapeutic standard for advanced gastric cancer, while limiting toxicity and preserving patients' quality of life, and could become the reference treatment to accompany the targeted therapies currently being developed for this disease.

The primary objective of this randomised phase III trial is to compare the progression-free survival on dual therapy with 5FU-oxaliplatin (FOLFOX protocol) with triple therapy with 5FU-oxaliplatin-docetaxel (TFOX protocol) in treatment of advanced forms of gastric or oesophagogastric junction adenocarcinoma. The secondary objectives are overall survival, the tumour response rate, toxicity, quality of life and the therapeutic index, defined as the ratio between the median progression-free survival and the febrile neutropenia rate.

ELIGIBILITY:
Inclusion Criteria:

* Gastric or gastro-oesophageal junction adenocarcinoma (all Siewert), histologically proven (on primary tumour or metastatic lesion),
* HER2 negative (positive HER2 status is defined by a positive IHC test of 3+ or IHC of 2+ with positive FISH)
* Metastatic or non-resectable (locally advanced) disease
* Disease measurable according to RECIST v1.1 criteria (at least one measurable lesion)
* No major surgical procedure during the 4 weeks prior to randomisation:
* Patient eligible for a 1st line of chemotherapy based on 5FU, folinic acid and oxaliplatin (FOLFOX) with or without docetaxel (TFOX)
* WHO: 0-1
* Age ≥ 18
* BMI > 18
* Life expectancy > 3 months
* PNN > 1500/mm3, platelets > 100,000/mm3, Hb > 10 g/dL
* AST, ALT ≤ 3.5 times the UNL, alkaline phosphatase < 6 times the UNL
* Bilirubin ≤ 1.5 times the UNL,
* Creatinine clearance according to Cockcroft and Gault formula > 50 mL/min
* Women of childbearing age must have a negative pregnancy test (β HCG) before starting treatment
* Women of childbearing age and men (who are in a sexual relationship with women of childbearing age) must agree to use effective contraception without interruption for the duration of the treatment and for 6 months after administration of the last dose of treatment
* Patient affiliated to a social security scheme
* Patient information and signature of informed consent form

Exclusion Criteria:

* Presence of cerebral or meningeal metastases
* Presence of > grade 2 neuropathy according to NCIC-CTC 4.0
* Known DPD deficiency
* QT/QTc interval > 450 msec for men and > 470 msec for women
* K+ < LNL, Mg2+ < LNL, Ca2+ < LNL
* Any known specific contraindication or allergy to the treatments used in the study (cf RCP Appendix 7)
* Chemotherapy or radio-chemotherapy in an adjuvant situation finished less than 12 months ago
* Prior chemotherapy including oxaliplatin (except for adjuvant chemotherapy)
* Prior chemotherapy including docetaxel
* Any progressive pathology not stabilised over the past 6 months: liver impairment, renal impairment, respiratory or cardiac failure
* HIV+ patients
* Radiotherapy during the 4 weeks prior to randomisation
* Other concomitant cancer or a history of cancer during the previous 5 years, with the exception of carcinoma in situ of the cervix or basal cell carcinoma or epidermoid cell carcinoma of the skin which is considered to be cured
* Patient already included in another clinical trial involving an experimental drug
* Pregnant or breastfeeding woman
* Persons in custody or under wardship
* Impossibility of undergoing medical monitoring during the trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 12 months after laste randomisation

SECONDARY OUTCOMES:
Overall survival Toxicity events (adverse events) according to NCI-CTC v4.0 | 12 months after laste randomisation
Objective response rate | 12 months after laste randomisation
Toxicity events according to NCI-CTC v4.0 | 12 months after laste randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Aziz ZAANAN, Study Chair — HEGP, Paris
Locations (133):
- France (131):
  - CH d'Abbeville, Abbeville
  - CHU Amiens-Picardie, Amiens
  - CHU d'Angers, Angers
  - Hôpital Privé D'Antony, Antony
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - CH d'Auxerre, Auxerre
  - CH de la Côte Basque, Bayonne
  - CH, Beauvais
  - Centre de Radiothérapie Pierre Curie, Beuvry
  - CH Germont et Gauthier, Béthune
  - Centre Hospitalier Germon Et Gauthier, Béthune
  - CH de Blois, Blois
  - Clinique Tivoli, Bordeaux
  - Institut Bergonie, Bordeaux
  - Polyclinique de Bordeaux Nord, Bordeaux
  - Polyclinique Saint Privat, Boujan-sur-Libron
  - CMCO Côte d'Opale, Boulogne-sur-Mer
  - Hôpital Duchenne, Boulogne-sur-Mer
  - Centre Hospitalier Fleyriat, Bourg-en-Bresse
  - Hôpital Pierre Oudot, Bourgoin
  - Centre Hospitalier Pierre Oudot, Bourgoin
  - CHU Côte de Nacre, Caen
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Médipôle de Savoie, Challes-les-Eaux
  - CH William Morey, Chalon-sur-Saône
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - CH Metropole Savoie, Chambéry
  - Hopital Prive Paul D Engine, Champigny-sur-Marne
  - Hopitaux de Chartres, Centre Hospitalier Louis Pasteur, Chartres
  - Centre Hospitalier Général, Châlons-en-Champagne
  - Centre Hospitalier de Cholet, Cholet
  - Hopital D Instruction Des Armées Percy, Clamart
  - Hopitaux civils de Colmar, Colmar
  - Clinique Saint Côme, Compiègne
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Clinique des Cèdres, Cornebarrieu
  - Groupe Hospitalier Du Sud de L'Oise, Creil
  - Hôpital Henri Mondor, Créteil
  - CHI, Créteil
  - Institut de Cancérologie de Bourgogne - GRRECC, Dijon
  - Centre Georges-François Leclerc, Dijon
  - CHU, Dijon
  - Centre Hospitalier de Dinan, Dinan
  - CHI Elbeuf-Louvier-Val de Reuil, Elbeuf
  - Centre Hospitalier Intercommunal Elbeuf-Louviers/Val de Reuil, Elbeuf
  - Hôpital Jacques Monod, Flers
  - CHI de Fréjus Saint-Raphaël, Fréjus
  - GHM Institut Daniel Hollard, Grenoble
  - Chu Albert Michallon, Grenoble
  - Hôpital privé Toulon/Hyères, Hyères
  - CHD Vendée, La Roche-sur-Yon
  - CHU Grenoble - Hôpital Albert Michallon, La Tronche
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Chu Claude Huriez, Lille
  - Clinique François Chénieux, Limoges
  - CHU Dupuytren, Limoges
  - CH Longjumeau, Longjumeau
  - Clinique de la Sauvegarde, Lyon
  - CHU de Lyon - Croix Rousse, Lyon
  - CH Saint Joseph - Saint Luc, Lyon
  - Centre Léon Berard, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hopital Saint Joseph -Saint Luc, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Centre Hospitalier Francois Quesnay, Mantes-la-Jolie
  - CHU La Timone, Marseille
  - Hôpital Nord, Marseille
  - Association Hopital Saint Joseph de Marseille, Marseille
  - Hôpital Européen, Marseille
  - CH, Meaux
  - Hopital Marc Jacquet, Melun
  - Centre Hospitalier, Montélimar
  - Ghi Le Raincy-Montfermeil, Montfermeil
  - Hôpital Monod, Montivilliers
  - Institut Régional du Cancer Montpellier, Montpellier
  - Chu de Nancy, Nancy
  - Hôpital privé du Confluent SAS, Nantes
  - Chu de Nantes, Nantes
  - CH Pierre Bérégovoy, Nevers
  - CH de Niort, Niort
  - CH Régional de la Source, Orléans
  - Hôpital de la source, Orléans
  - CHU Cochin, Paris
  - Croix Saint Simon, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Tenon, Paris
  - Centre Hospitalier Paris Saint Joseph, Paris
  - Groupe Hospitalier Pitié Salpêtrière, Paris
  - Hôpital Saint Louis, Paris
  - Institut Mutualiste Montsouris, Paris
  - Centre Hospitalier, Pau
  - Centre Hospitalier Saint Jean, Perpignan
  - Hôpital Haut Leveque, Pessac
  - Polyclinique Francheville, Périgueux
  - CHU Lyon Sud, Pierre-Bénite
  - Hôpital de la Milétrie, Poitiers
  - CH Annecy Genevois, Pringy
  - CHU Robert Debré, Reims
  - Institut Jean Godinot, Reims
  - Centre Hospitalier de Romans Sur Isere, Romans-sur-Isère
  - CHU Charles Nicolle, Rouen
  - Chi Poissy Saint Germain, Saint-Germain-en-Laye
  - Centre Hospitalier Prive Saint Gregoire, Saint-Grégoire
  - Clinique de L Union, Saint-Jean
  - Polyclinique Côte Basque, Saint-Jean-de-Luz
  - Centre Joliot Curie, Saint-Martin-Boulogne
  - Clinique Mutualiste de L Estuaire, Saint-Nazaire
  - CHU de Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez
  - Institut Lucien Neuwirth, Saint-Priest-en-Jarez
  - Plyclinique Saint Claude, Saint-Quentin
  - Clinique Trenel, Sainte-Colombe
  - Clinique Charcot, Sainte-Foy-lès-Lyon
  - Centre de cancérologie, Sarcelles
  - CH, Senlis
  - Centre Hospitalier de Soissons, Soissons
  - Centre Hospitalier de Saint Malo, St-Malo
  - Clinique de La Cote D Emeraude, St-Malo
  - Clinique Sainte Anne, Strasbourg
  - Centre Paul Strauss, Strasbourg
  - Les Hopitaux Universitaires de Strasbourg, Strasbourg
  - Hôpitaux du Leman, Thonon-les-Bains
  - Clinique Pasteur, Toulouse
  - Hôpital Trousseau, Tours
  - Centre Hospitalier de Troyes, Troyes
  - entre Hospitalier, Valenciennes
  - CHU Nancy-Brabois, Vandœuvre-lès-Nancy
  - Hôpital Privé de Villeneuve d'Asq, Villeneuve-d'Ascq
  - Centre Hospitalier Intercommunal, Villeneuve-Saint-Georges
  - Medipole Hopital Mutualiste Lyon Villeurbanne, Villeurbanne
  - HEGP, Paris, Île-de-France Region
- Martinique (2):
  - CHU de Fort de France, Fort-de-France
  - Chu Martinique, Fort-de-France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zaanan A, Samalin E, Aparicio T, Bouche O, Laurent-Puig P, Manfredi S, Michel P, Monterymard C, Moreau M, Rougier P, Tougeron D, Taieb J, Louvet C. Phase III randomized trial comparing 5-fluorouracil and oxaliplatin with or without docetaxel in first-line advanced gastric cancer chemotherapy (GASTFOX study). Dig Liver Dis. 2018 Apr;50(4):408-410. doi: 10.1016/j.dld.2018.01.119. Epub 2018 Mar 1. PMID 29409778
- [Derived] Zaanan A, Bouche O, de la Fouchardiere C, Le Malicot K, Pernot S, Louvet C, Artru P, Le Brun Ly V, Aldabbagh K, Khemissa-Akouz F, Lecomte T, Castanie H, Laly M, Botsen D, Roth G, Samalin E, Muller M, Breysacher G, Manfredi S, Phelip JM, Taieb J. TFOX versus FOLFOX in first-line treatment of patients with advanced HER2-negative gastric or gastro-oesophageal junction adenocarcinoma (PRODIGE 51- FFCD-GASTFOX): an open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2025 Jun;26(6):732-744. doi: 10.1016/S1470-2045(25)00130-5. Epub 2025 Apr 23. PMID 40286809